CLINICAL TRIAL: NCT00254202
Title: A Randomized, Double-blind, Placebo- and Active-controlled, Multicenter Study to Evaluate the Efficacy, Safety and Tolerability of Iloperidone in Schizophrenic Patients in Acute Exacerbation Followed by a Long-term Treatment Phase.
Brief Title: Efficacy and Safety of Iloperidone Compared With Placebo and Active Control in Subjects With Acute Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VYV-683-3101
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Atypical antipsychotic; Psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — iloperidone; ziprasidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Iloperidone (Experimental): Oral iloperidone
  Interventions: Drug: Iloperidone
- Ziprasidone (Active Comparator): Oral ziprasidone
  Interventions: Drug: Ziprasidone
- Placebo (Placebo Comparator): Oral placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Iloperidone
  Other Names: Fanapt®; VYV-683
  Arms: Iloperidone
Drug: Ziprasidone
  Arms: Ziprasidone
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and efficacy of iloperidone compared to placebo and an active comparator in the treatment of patients with schizophrenia in acute exacerbation.

DETAILED DESCRIPTION:
Schizophrenia is a severe mental illness affecting an estimated 1% of the world's population. Patients with schizophrenia suffer from productive symptoms (e.g., hallucinations and delusions), and deficit symptoms (e.g., a reduction or absence of normal behaviors or emotions). Other symptoms include a reduced ability to recall and learn new information.

Iloperidone is being development as a treatment for symptoms of schizophrenia. This trial will test the safety and efficacy of iloperidone in patients with an acute exacerbation of the disease.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia
* PANSS-T of at least 70 at screening and baseline

Exclusion Criteria:

* Clinically significant disease of the heart, kidneys, liver or gastrointestinal system
* DSM-IV diagnosis of psychiatric disorder other than schizophrenia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 593 (Actual)
Dates: Start 2005-11-18 (Actual); Primary Completion 2006-09-26 (Actual); Study Completion 2007-03-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (31):
  - Vanda Investigational Site, Little Rock, Arkansas
  - Vanda Investigational Site, Anaheim, California
  - Vanda Investigational Site, Cerritos, California
  - Vanda Investigational Site, Garden Grove, California
  - Vanda Investigational Site, Glendale, California
  - Vanda Investigational Site, Los Angeles, California
  - Vanda Investigational Site, National City, California
  - Vanda Investigational Site, Oceanside, California
  - Vanda Investigational Site, Paramount, California
  - Vanda Investigational Site, Pico Rivera, California
  - Vanda Investigational Site, San Diego, California
  - Vanda Investigational Site, Santa Ana, California
  - Vanda Investigational Site, Upland, California
  - Vanda Investigational Site, Bradenton, Florida
  - Vanda Investigational Site, Fort Lauderdale, Florida
  - Vanda Investigational Site, Maitland, Florida
  - Vanda Investigational Site, Atlanta, Georgia
  - Vanda Investigational Site, Augusta, Georgia
  - Vanda Investigational Site, Hoffman Estates, Illinois
  - Vanda Investigational Site, Lake Charles, Louisiana
  - Vanda Investigational Site, Rockville, Maryland
  - Vanda Investigational Site, Saint Charles, Missouri
  - Vanda Investigational Site, St Louis, Missouri
  - Vanda Investigational Site, Clementon, New Jersey
  - Vanda Investigational Site, Brooklyn, New York
  - Vanda Investigational Site, Cincinnati, Ohio
  - Vanda Investigational Site, Philadelphia, Pennsylvania
  - Vanda Investigational Site, Austin, Texas
  - Vanda Investigational Site, Houston, Texas
  - Vanda Investigational Site, Irving, Texas
  - Vanda Investigational Site, Richmond, Virginia
- India (9):
  - Vanda Investigational Site, Tirupati, Andhra Pradesh
  - Vanda Investigational Site, Ahmedabad, Gujarat
  - Vanda Investigational Site, Manipal, Karnataka
  - Vanda Investigational Site, Aurangabad, Maharashtra
  - Vanda Investigational Site, Pune, Maharashtra
  - Vanda Investigational Site, Jaipur, Rajasthan
  - Vanda Investgational Site, Chennai, Tamil Nadu
  - Vanda Investigational Site, Lucknow, Uttar Pradesh
  - Vanda Investigational Site, Chinawaltair, Visakha Patnam

REFERENCES:
- [Derived] Volpi S, Potkin SG, Malhotra AK, Licamele L, Lavedan C. Applicability of a genetic signature for enhanced iloperidone efficacy in the treatment of schizophrenia. J Clin Psychiatry. 2009 Jun;70(6):801-9. doi: 10.4088/jcp.08m04391. PMID 19573479

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Iloperidone | Ziprasidone | Placebo
Started (Randomized (excluding randomization errors)) | 295 | 149 | 149
Safety Population | 300 | 150 | 147
Completed | 193 | 98 | 90
Not Completed | 102 | 51 | 59

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iloperidone | Ziprasidone | Placebo | Total
Number analyzed (Participants) | 295 | 149 | 149 | 593
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (10.4) | 40.0 (9.9) | 40.7 (10.4) | 39.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 36 | 35 | 121
  Male | 245 | 113 | 114 | 472
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 2 | 0 | 1 | 3
  Asian | 25 | 12 | 15 | 52
  Black or African American | 147 | 76 | 76 | 299
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 2
  White | 111 | 51 | 46 | 208
  Other | 8 | 10 | 11 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Symptom Scale Total (PANSS-T) Score
Description: The PANSS is a 30-item scale developed to assess the severity of symptoms of schizophrenia. The PANSS items are divided into positive, negative, and general psychopathology factors. Items are rated on a scale of 1 (absent) to 7 (extremely severe). The PANSS-T score is the sum of scores for all 30 PANSS items (i.e., the sum of the three subscales), with a minimum score of 30 and a maximum score of 210. Higher scores indicate more severe symptoms. A negative change from baseline indicates improvement.
Time Frame: 4 weeks
Population: The modified Intent-to-Treat (ITT) population comprise all randomized patients who receive at least one dose of study medication in the short-term double-blind phase and for whom a baseline PANSS score measurement is obtained and at least one post-baseline PANSS score measurement is obtained while on study medication. For patients randomized in error at a second site after being randomized once, the data from the second site were excluded from analysis in the modified ITT population.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Iloperidone | Ziprasidone | Placebo
Number analyzed (Participants) | 283 | 144 | 140
score on a scale | -12.0 (1.03) | -12.3 (1.44) | -7.1 (1.48)

ADVERSE EVENTS:
Description: The safety analysis included patients who received 1 or more doses of study medication and 1 or more subsequent safety evaluations. To provide the most conservative assessment of safety, the 10 patients erroneously randomized twice, who received study drug at each site and met the safety criteria, were counted twice in the safety population.
Arm/Group | Iloperidone | Ziprasidone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/300 | 0/150 | 0/147
Serious Adverse Events (participants affected / at risk) | 2/300 | 2/150 | 5/147
Other Adverse Events (participants affected / at risk) | 221/300 | 118/150 | 86/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Iloperidone (N=300) | Ziprasidone (N=150) | Placebo (N=147)
Microcytic anemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 2 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 2
Schizophrenia (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Iloperidone (N=300) | Ziprasidone (N=150) | Placebo (N=147)
Dizziness (Nervous system disorders) | 51 | 20 | 11
Sedation (Nervous system disorders) | 38 | 41 | 12
Weight increased (Investigations) | 34 | 7 | 3
Dry mouth (Gastrointestinal disorders) | 26 | 11 | 1
Heart rate increased (Investigations) | 24 | 9 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 25 | 5 | 4
Tachycardia (Cardiac disorders) | 28 | 3 | 1
Extrapyramidal disorder (Nervous system disorders) | 10 | 14 | 3
Agitation (Psychiatric disorders) | 10 | 10 | 4
Orthostatic hypotension (Vascular disorders) | 21 | 0 | 3
Somnolence (Nervous system disorders) | 12 | 9 | 2
Restlessness (Psychiatric disorders) | 11 | 8 | 3
Anxiety (Psychiatric disorders) | 9 | 8 | 1
Akathisia (Nervous system disorders) | 4 | 11 | 0
Headache (Nervous system disorders) | 61 | 35 | 29
Nausea (Gastrointestinal disorders) | 29 | 21 | 13
Dyspepsia (Gastrointestinal disorders) | 24 | 15 | 15
Constipation (Gastrointestinal disorders) | 27 | 12 | 14
Vomiting (Gastrointestinal disorders) | 17 | 16 | 10
Diarrhoea (Gastrointestinal disorders) | 20 | 12 | 10
Fatigue (General disorders) | 16 | 9 | 7
Stomach discomfort (Gastrointestinal disorders) | 13 | 7 | 8
Toothache (Gastrointestinal disorders) | 14 | 6 | 8
Decreased appetite (Metabolism and nutrition disorders) | 4 | 6 | 8
Insomnia (Psychiatric disorders) | 14 | 10 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days